CLINICAL TRIAL: NCT00336739
Title: The Effect of Cinacalcet on Gastric Acid Output in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2455
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Gastric acidity determination; Calcium sensing receptor
MeSH Terms: interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cinacalcet

SUMMARY:
The purpose of this study is to determine whether cinacalcet will increase gastric acid secretion in healthy volunteers.

DETAILED DESCRIPTION:
The calcium sensing receptor (CaSR) was originally found on parathyroid and renal cells and more recently it has been identified on cells that regulate gastric acid secretion (G cells and parietal cells). However, its role in regulating acid secretion in humans is completely unknown and is of potential importance because an acid environment in the stomach enhances intestinal calcium absorption. In this pilot project, we will stimulate the CaSR with a CaSR-agonist called cinacalcet. Our hypothesis is that activation of the CaSR will in turn increase gastric acid production in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory men and postmenopausal women
* Age 45 to 70
* Avoid alcohol, antacids, H2 blockers, proton pump inhibitors, or antihistamines during the study.

Exclusion Criteria:

* Ionized Ca++ level <4.39 mg/dl or >5.02 mg/dl (normal reference range 4.18- 5.02).
* 24-hour UCa++ excretion >350 mg.
* Cr >1.3.
* AST/ALT values >10% beyond reference range.
* Hgb level <11.7 g/dl in women and <13.2 g/dl in men.
* MCV level >102 UM3.
* Basal acid output >5 mEq/h in men and >3.8 mEq/h in women.
* Basal acid output <1 mEq/h in men and <0.2 mEq/h in women.
* Age <45 or >70.
* Premenopausal or <1 year post-menopause.
* Individuals following vegan diets.
* Current EtOH abuse.
* Lidocaine allergy. Medications
* Antacids
* H2 blockers
* Proton pump inhibitors
* Carafate
* Anticholinergic agents (i.e. TCA)
* Cholinergic agents
* Antihistamines in the last 3 weeks
* Cogentin
* Adrenergic blockers
* Thiazide diuretics
* Antiplatelet drugs
* Oral and Inhaled Glucocorticoids
* Bisphosphonates
* Raloxifene, Tamoxifen
* Tobacco
* EtOH during study
* rPTH
* Calcitonin
* Ketoconazole/Itraconazole
* Calcitriol
* Paricalcitol
* Drisdol, Ergocalciferol
* Phosphate binders
* Anticoagulant
* Erythromycin
* Hormone replacement therapy except vaginal estrogen creams

Exclusion Diseases

* Achlorhydria
* Pernicious anemia
* Zollinger Ellison syndrome
* Congestive heart failure
* Esophageal strictures or motility problems
* History of a GI bleed
* Prior upper GI surgery
* Malabsorption
* History of GI malignancy
* GERD, gastritis, duodenitis
* Active peptic ulcer disease
* Gallbladder disease
* Liver disease
* Pancreatitis
* Current kidney stone
* Renal disease
* Current hypoparathyroidism or hyperparathyroidism
* Moderate to Severe coronary artery disease
* Aortic aneurysm
* Seizure disorder
* Current Arrhythmia

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Compare change in gastric acid output in response to an 11-day course of daily cinacalcet or placebo in subjects on a fixed protein metabolic diet. | 11 days

SECONDARY OUTCOMES:
Compare serum gastrin levels in subjects before and after an 11-day course of cinacalcet or placebo and on a fixed protein metabolic diet. | 11 days
Compare 24-hour urinary calcium excretion before and after an 11-day course of cinacalcet or placebo and on a fixed protein metabolic diet. | 11 days
Compare serum IGF-1 levels before and after an 11-day course of cinacalcet or placebo and on a fixed protein metabolic diet. | 11 days
Compare change in urinary magnesium excretion in response to an 11-day course of daily cinacalcet or placebo in subjects on a fixed protein metabolic diet. | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Human Nutrition Research Center on Aging at Tufts University
Locations (1):
- Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ceglia L, Harris SS, Rasmussen HM, Dawson-Hughes B. Activation of the calcium sensing receptor stimulates gastrin and gastric acid secretion in healthy participants. Osteoporos Int. 2009 Jan;20(1):71-8. doi: 10.1007/s00198-008-0637-8. Epub 2008 Jun 7. PMID 18536954